CLINICAL TRIAL: NCT02585115
Title: Is a First Void Urine Sample as Accurate as a Midstream Urine Sample in Diagnosing Urinary Tract Infections With a Point-Of-Care-Test Method in Adult, Symptomatic, Non-pregnant Women in General Practice?
Brief Title: Diagnostic Accuracy of Point of Care Test of First Voided Urine Compared to Midstream Voided Urine in Primary Care
Status: Completed | Type: Observational
Sponsor: University of Copenhagen (Other)
Responsible Party: Principal Investigator, Pernille Brunsgaard, Medical Student, University of Copenhagen
Other Study IDs: UCCAREWP4Samples
Record Dates: First submitted 2015-10-05; First posted 2015-10-23 (Estimated); Last update posted 2016-10-06 (Estimated); Status verified 2016-10

CONDITIONS: Urinary Tract Infections
MeSH Terms: conditions — Urinary Tract Infections

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Non-pregnant women with symptoms: Non-pregnant women with one or more symptoms of UTI. All women will make a paired urine sample (first void and midstream void) of the same urine sample.

SUMMARY:
The aim of this study is to determine if sampling technique of urine affects diagnostic modalities in primary care. Furthermore it aims to determine if there is difference in the accuracy of the point-of-care test, when the urine sample is stored at room-temperature and analyzed later in the day.

DETAILED DESCRIPTION:
125 patients with one or more symptoms of urinary tract infections, contacting their GP, are asked to make 2 urine samples from the same void. The patient is asked to void firstly in one cup, approximately 10-20 ml., then stop voiding. Then the patient is asked to void the rest into a second cup. This way there is collected both a first-void and a midstream-void from the same patient and the same void.

All the samples are analyzes using urine-dipstick, microscopy and point of care test urine culture. The urine of the midstream void is sent to a Microbiology lab for analyzes as well. Furthermore the test are analyzes again after 1 and 4 hours.

ELIGIBILITY:
Inclusion Criteria:

* Symptoms of urinary tract infection

Exclusion Criteria:

* Men
* Pregnancy
* Children
* Unable to understand the verbal and written guide

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Non-pregnant adult women with symptoms of UTI all included in General Practice.
Sampling Method: Non-Probability Sample
Enrollment: 117 (Actual)
Dates: Start 2015-10; Primary Completion 2016-07 (Actual); Study Completion 2016-07 (Actual)

PRIMARY OUTCOMES:
Difference in accuracy of POC urine culture on first-void urine compared to mid-stream urine wtih mid-stream urine microbiological culture as a reference | 1 year
Difference in accuracy from 0 hours to 4 hours of the POCT Flexicult ID in the most precise of the above techniques. | 1 year

SECONDARY OUTCOMES:
Proportion of false-positive cultures after 0 hours at room temperature with first-void urine compared to mid-stream urine when using a urin-dipstick | 1 year
Proportion of false-positive cultures after 0 hours at room temperature with first-void urine compared to mid-stream urine when using microscopy | 1 year
Proportion of false-positive cultures after 1 hours at room temperature with first-void urine compared to mid-stream urine when using a urin-dipstick | 1 year
Proportion of false-positive cultures after 1 hours at room temperature with first-void urine compared to mid-stream urine when using microscopy | 1 year
Proportion of false-positive cultures after 4 hours at room temperature with first-void urine compared to mid-stream urine when using a urin-dipstick | 1 year
Proportion of false-positive cultures after 4 hours at room temperature with first-void urine compared to mid-stream urine when using microscopy | 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Pernille Brunsgaard, med.stud., Principal Investigator — Research Unit of General Practice, Odense
Locations (1):
- Vesterbro Lægehus, Copenhagen, Denmark